CLINICAL TRIAL: NCT02976389
Title: Southern California Nutrition Incentive Program
Acronym: SCNIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The California Endowment (Other); The Ecology Center (Unknown); Center for Good Food Purchasing (Unknown); Northgate Gonzalez Markets (Unknown); Latino Health Access (Unknown); California Department of Health Services (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kay Rhee, Associate Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-70025-25247
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Food Insecurity
Keywords: Supplemental Nutrition Assistance Program; Food insecurity; fruit and vegetable; healthy diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- $40/month (Experimental): Financial incentives: Participants will be randomized to receive $40/month in incentive dollars for the purchase of SNAP eligible fruits and vegetables. Purchasing behaviors will be tracked.
  Interventions: Other: Financial Incentive: High
- $20/month (Active Comparator): Financial Incentives: Participants will be randomized to receive $20/month in incentive dollars for the purchase of SNAP eligible fruits and vegetables. Purchasing behaviors will be tracked.
  Interventions: Other: Financial Incentive: Middle
- $10/month (Active Comparator): Financial Incentives: Participants will be randomized to receive $10/month in incentive dollars for the purchase of SNAP eligible fruits and vegetables. Purchasing behaviors will be tracked.
  Interventions: Other: Financial Incentive: Low

INTERVENTIONS:
Other: Financial Incentive: High — dlParticipants in this group will receive an additional $40/month to use towards the purchase of SNAP eligible fruits and vegetables. They will be able to access these dollars through an electronic wallet (e-wallet) that is tied to their customer loyalty card. They will also have access to the fruit and vegetable promotions that include discount pricing and SNAP-Ed programming (e.g., in-store cooking classes, tours, and healthy food self-labeling system) to educate and support the purchasing behaviors of SNAP-eligible families.
  Other Names: Mas Fresco
  Arms: $40/month
Other: Financial Incentive: Middle — Participants in this group will receive an additional $20/month to use towards the purchase of SNAP eligible fruits and vegetables. They will be able to access these dollars through an electronic wallet (e-wallet) that is tied to their customer loyalty card. They will also have access to the fruit and vegetable promotions that include discount pricing and SNAP-Ed programming (e.g., in-store cooking classes, tours, and healthy food self-labeling system) to educate and support the purchasing behaviors of SNAP-eligible families.
  Other Names: Mas Fresco
  Arms: $20/month
Other: Financial Incentive: Low — Participants in this group will receive an additional $10/month to use towards the purchase of SNAP eligible fruits and vegetables. They will be able to access these dollars through an electronic wallet (e-wallet) that is tied to their customer loyalty card. They will also have access to the fruit and vegetable promotions that include discount pricing and SNAP-Ed programming (e.g., in-store cooking classes, tours, and healthy food self-labeling system) to educate and support the purchasing behaviors of SNAP-eligible families.
  Other Names: Mas Fresco
  Arms: $10/month

SUMMARY:
The specific aims of this proposal are to implement SCNIP in 6 Northgate Gonzalez Markets across San Diego, Orange and LA counties (2 in each county), and determine which level of financial incentive rebate (specifically, $10/month, $20/month, or $40/month) optimally increases the purchase and consumption of SNAP eligible fruits and vegetables.

DETAILED DESCRIPTION:
The University of California San Diego (UCSD) Center for Community Health, in collaboration with Northgate Gonzalez Markets and its regional partners, will implement a Food Insecurity Nutrition Incentive program in Los Angeles, Orange and San Diego Counties - the Southern California Nutrition Incentive Program (SCNIP). This program will develop, implement and evaluate a multi-tiered model that will enable low-income, SNAP-eligible consumers to make healthier food choices and purchase more fruits and vegetables. This model will include: tier 1) an innovative fruit and vegetable financial incentive rebate program that utilizes the consumer's Northgate Gonzalez Market customer loyalty card, electronic benefit transfer (EBT) card, and electronic wallet (e-wallet); tier 2) fruit and vegetable promotions that include discount pricing; and tier 3) SNAP-Ed programming (e.g., in-store cooking classes, tours, and healthy food self-labeling system) to educate and support the purchasing behaviors of SNAP-eligible families. Through the use of the customer loyalty card, EBT card, and e-wallet, the rebate program will be able to track the purchase of SCNIP eligible fruits and vegetables and provide a rebate at the point-of-sale that can be used to purchase additional fruits and vegetables, thus increasing the purchasing power of SNAP-eligible families for healthy food options. Earned and dispensed rebate dollars will be stored on the e-wallet enabling the tracking of purchasing behaviors and dollars spent on healthy fruits and vegetables in this program. With this data, we will be able to determine what level of financial incentive rebate ($10/month, $20/month, or $40/month) (tier 1) optimally increased SNAP families' per capita spending on fruits and vegetables in conjunction with the fruit and vegetable promotions (tier 2) and nutrition education activities (tier 3).

ELIGIBILITY:
Inclusion Criteria:

* Northgate Gonzalez Market customer who currently receives SNAP benefits and has a valid EBT card
* 18 years of age or older
* Speaks and reads in English or Spanish
* Shops at the selected Northgate Gonzalez Market regularly, at least two times per month

Exclusion Criteria:

* Does not receive SNAP benefits
* Unable to complete surveys in English or Spanish
* Another immediate family member living in the same household is already recruited into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3780 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dollars spent on Fruits and Vegetables | 1 year
  Total amount of incentive dollars spent on Fruits and Vegetables per month
Quantity of Fruits and Vegetables | 1 year
  total quantity of fruits and vegetables purchased per month with incentive dollars

SECONDARY OUTCOMES:
Dietary intake | 1 year
  Change in self-reported fruit and vegetable consumption during the intervention
Six-item short form of the Food Security Survey Module | 1 year
  Change in food insecurity score at the end of the intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared with USDA on a quarterly basis. Data will include number of participants recruited, amount of incentive dollars used. USDA will determine when this data will be released